**Clinical Study Report Appendix 12.1.9** 

Drug Substance Acalabrutinib (ACP-196)

Study Code ACE-LY-005

# Appendix 12.1.9 Documentation of Statistical Methods and Supporting Statistical Analysis

Version 1.00 dated: 17 January 2020

**Protocol Number: ACE-LY-005** 

Protocol Title: A Phase 1b/2 Proof-of-Concept Study of the Combination of

ACP-196 and Pembrolizumab in Subjects with Hematologic

**Malignancies** 

Version: 1.00

Version date: 17 January 2020

The undersigned have reviewed this plan and find it to be consistent with the requirements of the protocol as it applies to their respective areas



# CONFIDENTIAL

This document (and all copies thereof) is the property of Acerta Pharma and contains valuable trade secrets and confidential information, including proprietary technical and business information. By accepting this document, you agree that the Confidential Information contained herein will not be disclosed to others without prior written authorization from Acerta Pharma and shall only be used for the purposes intended by the document.


# **Statistical Analysis Plan**

A Phase 1b/2 Proof-of-Concept Study of the Combination of ACP-196 and Pembrolizumab in Subjects with Hematologic Malignancies

**Protocol Number: ACE-LY-005** 

Version: 1.00

Date:17 January 2020

Study Statistician: PPD

Confidential Acerta Pharma 


# **TABLE OF CONTENTS**

| Table | e of C | contents | | 2 |
|---|---|---|---|---|
| Table | e of A | bbrevia | tions | 4 |
| 1 | INTE | RODUC | TION | 6 |
| 2 | OBJECTIVES | | | |
| | 2.1 | | y Objectives | |
| | 2.2 | | dary Objectives | |
| | 2.3 | Explora | atory Objectives: | 6 |
| 3 | STU | DY OVE | ERVIEW | 6 |
| | 3.1 | Study I | Design | 6 |
| | 3.2 | | e Size | |
| 4 | CTLI | רא באור | DPOINTS | 10 |
| 4 | 4.1 | | Endpoints | |
| | 4.1 | - | y Endpoints | |
| | | | Biomarker Analysis | |
| | | | • | |
| 5 | HYP | HYPOTHESES AND MULTIPLICITY14 | | |
| 6 | ANALYSIS SUBSETS | | | |
| | 6.1 | | ated Population | |
| | 6.2 | Efficac | y-evaluable Population | 14 |
| 7 | INTE | ERIM AN | IALYSIS | 14 |
| 8 | MIS | SING VA | ALUES | 14 |
| 9 | STA | TISTICA | AL METHODS OF ANALYSIS | 15 |
| | 9.1 General Principles | | | |
| | 9.2 | Subjec | t Accountability | 16 |
| | 9.3 Important Protocol Deviations | | | |
| | 9.4 | Baselir | ne Data | 17 |
| | | 9.4.1 | Demographics | 17 |
| | | 9.4.2 | Baseline Characteristics | 17 |
| | 9.5 | Treatm | ent and Medications | 17 |
| | | 9.5.1 | Prior Anticancer Therapies | 17 |
| | | 9.5.2 | Prior and Concomitant Medications Received for Indications Other than MCL | 18 |
| | | 9.5.3 | Exposure to Study Drug | |
| | 9.6 | Analys | es of Efficacy Endpoints | 18 |


| | 9.6.1 | Response Rate | 18 |
|---|---|---|---|
| | 9.6.2 | Duration of Response | 19 |
| | 9.6.3 | Progression-free Survival | 19 |
| | 9.6.4 | Time to Next Treatment | 20 |
| | 9.6.5 | Overall Survival | 20 |
| | 9.6.6 | Analysis Methods | 20 |
| 9.7 | Analys | es Safety Endpoints | 21 |
| | 9.7.1 | Adverse Events | 21 |
| | 9.7.2 | Laboratory Test Results | 21 |
| | 9.7.3 | Vital Signs | 22 |
| | 9.7.4 | ECOG Performance Status | 22 |
| | 9.7.5 | Physical Examinations | 22 |
| СНА | NGES F | FROM PROTOCOL-SPECIFIED ANALYSES | 22 |
| LITE | RATUR | E CITATIONS / REFERENCES | 22 |
| APP | ENDICE | ES | 24 |
| 12.1 Study day | | | |
| 12.2 | Censor | ring Rules for Duration of Response | 24 |
| | 12.4 Censoring Rules for Overall Survival26 | | |
| | CHA<br>LITE<br>APP<br>12.1<br>12.2<br>12.3 | 9.6.2<br>9.6.3<br>9.6.4<br>9.6.5<br>9.6.6<br>9.7 Analys<br>9.7.1<br>9.7.2<br>9.7.3<br>9.7.4<br>9.7.5<br>CHANGES F<br>LITERATUR<br>APPENDICE<br>12.1 Study of<br>12.2 Censor<br>12.3 Censor | 9.6.2 Duration of Response 9.6.3 Progression-free Survival 9.6.4 Time to Next Treatment 9.6.5 Overall Survival 9.6.6 Analysis Methods 9.7 Analyses Safety Endpoints 9.7.1 Adverse Events 9.7.2 Laboratory Test Results 9.7.3 Vital Signs 9.7.4 ECOG Performance Status. 9.7.5 Physical Examinations CHANGES FROM PROTOCOL-SPECIFIED ANALYSES LITERATURE CITATIONS / REFERENCES APPENDICES 12.1 Study day 12.2 Censoring Rules for Duration of Response 12.3 Censoring Rules for Progression-free Survival |


# **TABLE OF ABBREVIATIONS**

ACP-196 acalabrutinib

AE(s) adverse event(s)

ATC anatomical therapeutic chemical

BID twice per day

CI confidence interval

CLL chronic lymphocytic leukemia

CR complete response **CSR** clinical study report

CT computed tomography

**CTCAE** Common Terminology Criteria for Adverse Events

**DLBCL** diffuse large B-cell lymphoma

DLT dose-limiting toxicity DOR duration of response **ECG** electrocardiogram

**ECOG** Eastern Cooperative Oncology Group

eCRF electronic case report form **EDC** electronic data capturing

**EORTC** European Organisation for Research and Treatment of Cancer

FL follicular lymphoma **GCB** germinal center B-cell

**IPD** important protocol deviation

MCL mantle cell lymphoma

MedDRA Medical Dictionary for Regulatory Activities

MF myelofibrosis

MM multiple myeloma

NCI National Cancer Institute

ORR overall response rate

OS overall survival

PDprogressive disease PDpharmacodynamics

**PFS** progression-free survival

PK pharmacokinetics PR partial response

**Statistical Analysis Plan** 


PT preferred term

SAE(s) serious adverse event(s) SAP statistical analysis plan

stable disease SD

SD standard deviation

SLL small lymphocytic lymphoma

TEAE(s) treatment-emergent adverse events

US **United States** 

WHO World Health Organization

WM Waldenström macroglobulinemia


### 1 INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide details of the planned statistical analyses that have been outlined within Protocol Amendment 6 for Study ACE-LY-005, which is entitled "A Phase 1b/2 Proof-of-Concept Study of the Combination of ACP-196 and Pembrolizumab in Subjects with Hematologic Malignancies" dated 14 March 2019. Any changes to the methods described in the final SAP will be documented in the clinical study report (CSR). Hereafter, acalabrutinb (a generic name for ACP-196) will be used in place of ACP-196 in this document.

Separate reports will be generated for pharmacokinetic (PK) and pharmacodynamics (PD) data.

# **OBJECTIVES**

### 2.1 **Primary Objectives**

To characterize the safety profile of acalabrutinib and pembrolizumab in subjects with hematologic malignancies.

### Secondary Objectives 2.2

To evaluate the activity of acalabrutinib and pembrolizumab as measured by response rate, duration of response, progression-free survival, overall survival, and time to next treatment.

### 2.3 **Exploratory Objectives:**



# STUDY OVERVIEW

# 3.1 Study Design

This is a Phase 1b/2, open-label, nonrandomized study that will be conducted in 2 stages. In the first stage, Part 1 of the study will determine the safety and preliminary

Acerta Pharma 

Statistical Analysis Plan


efficacy of acalabrutinib and pembrolizumab in a limited group of B-cell malignancies. In the second stage, Part 2 allows for possible expansion cohorts into a wider range of Bcell malignancies, and Part 3 (enrolled concurrently with Part 2) will evaluate the combination in subjects with myelofibrosis (MF).

# Part 1

Six subjects will be enrolled to receive acalabrutinib in combination with pembrolizumab. If the combination is safe with ≤ 1 dose-limiting toxicity (DLT) (6-week observation period) in the first 6 subjects, the cohort will be expanded up to 24 subjects to obtain additional safety information and to assess the efficacy of the combination.

Part 1 of the study will include adult subjects with the following disease types:

- Non-GCB diffused large B-cell lymphoma (DLBCL)
- Follicular lymphoma (FL)
- Chronic lymphocytic leukemia (CLL)/Small lymphocytic lymphoma (SLL)

# Part 2

Part 2 consists of expansion groups of up to 30 subjects per histology provided the safety and efficacy results from Part 1 of the study indicate that further evaluation of the combination is warranted. The possible expansion groups for Part 2 could include adult subjects with the following disease types:

- Non-GCB DLBCL
- GCB DLBCL
- Richter syndrome (RS)
- Mantel cell lymphoma (MCL)
- Non-Hodgkin lymphoma (iNHL)
  - o FL
  - Waldenström Macroglobulinemia (WM)
  - o CLL/SLL
- Multiple Myeloma (MM)
- Other B-cell malignancy (including but not limited to: Hodgkin's lymphoma, Burkitt lymphoma, marginal zone lymphomas, mediastinal large B-cell lymphoma, and hairy cell leukemia)

Under Amendment 3 of this protocol, subjects with MCL or iNHL (including FL, WM, and CLL/SLL) are no longer enrolled. Under Amendment 4, subjects with RS are no longer enrolled.

Statistical Analysis Plan


# Part 3

Part 3 includes up to 30 subjects with primary MF, post-polycythemia vera MF, or postessential thrombocythemia MF with thrombocytopenia or anemia. Part 3 will run in parallel with Part 2. Subjects with MF will receive a run-in of 6 weeks of acalabrutinib alone.

Subjects who are demonstrating a clinically meaningful response, in the opinion of the investigator, may continue on acalabrutinib monotherapy; those who are not will be treated with combination therapy with acalabrutinib and pembrolizumab.

In Part 3, safety and response data will be reviewed after the initial 12 subjects have completed 24 weeks of treatment (i.e., the Week 25 visit) or have discontinued treatment before Week 25. The first 12 subjects will be evaluated regardless of the length of treatment with acalabrutinib alone or in combination with pembrolizumab. If < 2 subjects who received acalabrutinib monotherapy or the combination with pembrolizumab have achieved a response of "clinical improvement" or better. the MF group will not be expanded. The decision to expand the study is multifactorial and will take into consideration the nature and quality of response, safety, and evolving competitive landscape. If the safety and response data indicate that further evaluation is warranted, up to 18 additional subjects with MF (for a total of up to 30 subjects) will be treated on the same adaptive regimen as was given to the first 12 subjects.

Under Amendment 3 of this protocol, Part 3 is closed to enrollment.

# **All Parts**

Treatment with acalabrutinib may be continued until disease progression or an unacceptable drug-related toxicity occurs as defined in the protocol. Treatment with acalabrutinib can continue until the end of trial, defined as 48 months after the last subject is enrolled.

Subjects who are still on treatment at the end of the study and deriving clinical benefit from acalabrutinib treatment may be eligible to enroll in a separate rollover study. Treatment with pembrolizumab may continue for 24 months (103 weeks) from first dose of pembrolizumab, provided subjects are tolerating the drug and not progressing. In addition, pembrolizumab treatment can end for subjects with confirmed complete remission (CR) (or stringent complete remission [sCR] for MM) if treatment has been

Acerta Pharma 

**Statistical Analysis Plan** 


administered for at least 24 weeks and 2 doses of pembrolizumab have been administered after confirmation of CR/sCR. Subjects who have confirmed progressive disease will come off treatment. Note: If there is uncertainty regarding whether there is cancer progression, the subject may continue study treatment and remain under close observation (e.g., evaluated at 4- to 8-week intervals) pending confirmation of progression. In particular, transient worsening of disease during temporary interruption of study therapy (eg, for drug related toxicity or intercurrent illness) may not indicate disease progression. In such circumstances, and if medically appropriate, subjects may resume therapy and relevant clinical, laboratory, and/or radiographic assessments should be done to document whether tumor control can be maintained or whether actual disease progression has occurred.

All subjects will have bone marrow biopsy, hematology, chemistry, thyroid, and urinalysis safety panels performed at screening. Once dosing commences (Day 1), all subjects will be evaluated for safety, including serum chemistry, hematology, and thyroid function tests, once weekly for the first 8 weeks, followed by a Week 10 visit and then every 3 weeks thereafter (every 6 weeks thereafter for thyroid function tests) through Week 103. For subjects who discontinue pembrolizumab at Week 103, the Week 103 visit will be followed by Week 106 and Week 109 visits, at which time, the investigator will determine eligibility to continue single-agent acalabrutinib treatment. Subjects remaining on study treatment after Week 103 will have a Week 103 and Week 115 visit, and then visits for safety and tumor response assessments every 24 weeks starting at Week 127 through 3 years (for subjects with CLL/SLL histologies) or 5 years (for subjects with non-CLL/SLL histologies [i.e., DLBCL/Hodgkin lymphoma]), and then every 52 weeks thereafter (all histologies).

Subjects who permanently discontinue pembrolizumab at any time during study participation must have a minimum of 2 consecutive study visits, 3 weeks apart, after the last dose of pembrolizumab for safety evaluation. The study visits will be scheduled as follows:

- For all subjects except MM and CLL subjects
- If a subject discontinued pembrolizumab prior to completing 37 weeks on study and is on acalabrutinib alone, study visits will be held every 3 weeks until Week 37. After Week 37, study visits will be held every 12 weeks.

Acerta Pharma 

Statistical Analysis Plan


 If a subject discontinued pembrolizumab after completing 37 weeks on study and is on acalabrutinib alone, 2 consecutive study visits will be held 3 weeks apart (eg, Week 40 and 43), after which study visits will be held every 12 weeks.

 It is acknowledged that the discontinuation timepoint of pembrolizumab (if applicable) is unique per subject. To synchronize the every 12-week study visit schedule with the radiologic tumor assessment schedule, the first 2 study visits after pembrolizumab discontinuation should be 3 and 6 weeks after pembrolizumab discontinuation and then scheduled to align with the nearest radiological timepoint.

# For CLL subjects

- If a subject discontinued pembrolizumab prior to completing 37 weeks on study and is on acalabrutinib alone, study visits will be held every 3 weeks until Week 37. After Week 37, study visits will be held every 12 weeks.
- o If a subject discontinued pembrolizumab after completing 37 weeks on study and is on acalabrutinib alone, study visits will be held every 12 weeks.
- It is acknowledged that the discontinuation timepoint of pembrolizumab (if applicable) is unique per subject. To synchronize the every 12-week study visit schedule with the radiologic tumor assessment schedule, the first study visit should be scheduled to align with the nearest radiological timepoint. In addition, subjects who permanently discontinue pembrolizumab for any reason (eg, pembrolizumab toxicity, AE, or completing the 103-week course of pembrolizumab) and remain on acalabrutinib alone at any time during study participation must have a thyroid test done every 6 weeks for 6 months after pembrolizumab discontinuation. Thyroid testing may be discontinued at 6 months if 1) testing that was performed at 6 months was normal and 2) testing that was performed 6 weeks prior to the 6-month timepoint was normal (for a total of 2 consecutive normal test results). Otherwise, thyroid testing will continue as scheduled until 2 consecutive normal test results.

Refer to protocol Appendix 5 and Appendix 6 for a comprehensive list of study assessments and their timing.

Acerta Pharma 

Statistical Analysis Plan


# 3.2 Sample Size

In Part 1 (dose-limiting toxicity [DLT] review), enrollment of 6 subjects for DLT review is consistent with sample sizes used in oncology studies for determination of maximum toxicity dose (MTD). The trial employs the standard National Cancer Institute definition of MTD (dose associated with DLT in < 33.3% of subjects). Provided  $\leq$  1 DLT occurs during the DLT review, then expansion will occur in Part 1 to include up to 24 subjects in a select group of histologies. The safety and preliminary efficacy results from Part 1 will be used to determine opening Part 2 and Part 3 of the protocol.

In Part 2 (expansion groups), enrollment of 30 subjects offers the opportunity to determine if there is sufficient antitumor activity to warrant further development in the selected tumor types. An ORR of  $\geq$  20% is considered the minimum value of potential interest in each of the selected indications. If < 2 subjects per cohort experience an objective response, the probability is > 0.90 that an ORR of ≥ 20% will be excluded for that cancer. If 2 subjects in a group experience an objective response, the upper bound of a 1-sided exact binomial 90% CI = 16.8%.

In Part 3, safety and response data will be reviewed after the initial 12 subjects have completed 24 weeks of treatment (ie, the Week 25 visit) or have discontinued treatment before Week 25. The first 12 subjects will be evaluated regardless of the length of treatment with acalabrutinib alone or in combination with pembrolizumab. If < 2 subjects who received acalabrutinib monotherapy or the combination with pembrolizumab have achieved a response of "clinical improvement" or better, the myelofibrosis (MF) group will not be expanded. The decision to expand the study is multifactorial and needs to take into consideration the nature and quality of response, safety, and evolving competitive landscape. If the safety and response data indicate that further evaluation is warranted, up to 18 additional subjects with MF (for a total of up to 30 subjects) will be treated on the same adaptive regimen as was given to the first 12 subjects.

Table 3-1 shows the 2-sided exact 90% binomial CIs on the true response rate for the range of all possible values for the observed response rate in the initial group of 12 subjects.

Table 1. Two-Sided Exact 90% Cls for Response Rate in Initial Group in Part 3 (N=12)

Acerta Pharma 


| D | n Response Rate, % | 90%CI | |
|--------------|--------------------|-------------|-------------|
| Responses, n | | Lower Bound | Upper Bound |
| 0 | 0% | 0% | 22% |
| 1 | 8% | 0% | 34% |
| 2 | 17% | 3% | 44% |
| 3 | 25% | 7% | 53% |
| 4 | 33% | 12% | 61% |
| 5 | 42% | 18% | 68% |
| 6 | 50% | 25% | 75% |
| 7 | 58% | 32% | 82% |
| 8 | 67% | 39% | 88% |
| 9 | 75% | 47% | 93% |
| 10 | 83% | 56% | 97% |
| 11 | 92% | 66% | 100% |
| 12 | 100% | 78% | 100% |

Abbreviation: CI = confidence interval.

If the MF group is expanded, enrollment of 30 subjects offers the opportunity to determine if there is sufficient antitumor activity to warrant further development in MF. A response rate (clinical improvement, PR, or CR) of  $\geq$  25% within the sample size of 30 subjects with MF is considered the minimum value of potential interest in this highly unmet medical need population of MF patients with thrombocytopenia or anemia. To reject the null hypothesis of response rate  $\leq 5\%$  in favor of an alternative hypothesis that the response rate is  $\geq$  25%, 30 subjects will preserve approximately 90% power to detect the difference at a 0.05 level of significance by 1-sided exact test for single proportion. Considering the planned expansion cohort size of 30 subjects, Table 3-2 shows the 2-sided exact 90% binomial CIs on the true response rate for the range of all possible values for the observed response rate.

Acerta Pharma 


Table 3-2. Two-Sided Exact 90% CIs for Response Rate in Expansion Cohorts in Part 2 and Part 3 (N=30)

| D | Dannana Data N | 90%CI | |
|--------------|------------------|-------------|-------------|
| Responses, n | Response Rate, % | Lower Bound | Upper Bound |
| 0 | 0% | 0% | 10% |
| 1 | 3% | 0% | 15% |
| 2 | 7% | 1% | 20% |
| 3 | 10% | 3% | 24% |
| 4 | 13% | 5% | 28% |
| 5 | 17% | 7% | 32% |
| 6 | 20% | 9% | 36% |
| 7 | 23% | 11% | 39% |
| 8 | 27% | 14% | 43% |
| 9 | 30% | 17% | 47% |
| 10 | 33% | 19% | 50% |
| 11 | 37% | 22% | 53% |
| 12 | 40% | 25% | 57% |
| 13 | 43% | 28% | 60% |
| 14 | 47% | 31% | 63% |
| 15 | 50% | 34% | 66% |
| 16 | 53% | 37% | 69% |
| 17 | 57% | 40% | 72% |
| 18 | 60% | 43% | 75% |
| 19 | 63% | 47% | 78% |
| 20 | 67% | 50% | 81% |
| 21 | 70% | 53% | 83% |
| 22 | 73% | 57% | 86% |
| 23 | 77% | 61% | 89% |
| 24 | 80% | 64% | 91% |
| 25 | 83% | 68% | 93% |
| 26 | 87% | 72% | 95% |
| 27 | 90% | 76% | 97% |
| 28 | 93% | 80% | 99% |
| 29 | 97% | 85% | 100% |
| 30 | 100% | 90% | 100% |

Abbreviation: CI=confidence interval.

# **STUDY ENDPOINTS**

### 4.1 **Safety Endpoints**

- Frequency and severity of treatment-emergent AEs/SAEs.
- Relationship of AEs to study drug (eg, either acalabrutinib, pembrolizumab, or both).
- Change of laboratory parameters from baseline over time.
- Vital sign assessments, ECGs, and physical examinations


### 4.2 **Efficacy Endpoints**

- Response rate
- **Duration of response**
- Progression-free survival
- Time-to-next treatment
- Overall survival

### 4.3 PD or Biomarker Analysis

Additional PD and biomarker analyses may be performed, as deemed appropriate.

### HYPOTHESES AND MULTIPLICITY 5

No formal statistical hypothesis will be tested. The clinical hypothesis is that acalabrutinib and pembrolizumab is safe and effective in subjects with hematologic malignancies.

# **ANALYSIS SUBSETS**

### 6.1 **All Treated Population**

The safety analyses and primary efficacy analyses will be performed on the All-treated population, defined as all enrolled subjects who receive ≥1 dose of any study drug (either acalabrutinib or pembrolizumab).

### 6.2 **Efficacy-evaluable Population**

All subjects in the All-treated population who have ≥ 1 evaluable response assessment after the first dose of study drug (either acalabrutinib or pembrolizumab). Sensitivity analyses for efficacy will be carried out on the Efficacy-evaluable population.

# **INTERIM ANALYSIS**

No formal interim analysis was planned.

### **MISSING VALUES** 8

Statistical Analysis Plan


No imputation of values for missing data will be performed except that missing or partial start and end dates for AEs and concomitant medication will be imputed according to prespecified, conservative imputation rules. Subjects lost to follow-up (or drop out) will be included in statistical analyses to the point of their last evaluation.

Imputation of partial dates will be made for AE onset and stop dates, start and end dates of concomitant medication, start date of subsequent anticancer therapy, date of initial diagnosis and death date. If dates are completely missing, no imputation will be made. For any partial date with missing year, no imputation will be made.

The general rule for imputation is:

- If only day is missing, then the 15<sup>th</sup> of the month will be used.
- If only year is present, then June 30<sup>th</sup> will be used.

If such imputation date for initial diagnosis is on or after date of first dose, the date of first dose – 1 will be used. If such imputed date for subsequent anticancer therapies is before date of last dose, the date of last dose + 1 will be used.

If the imputed date is for an AE start date and is in the same year and month as the first dose date but before the first dose date, then the first dose date will be used, or if the imputed AE start date is after the AE end date, then the AE end date will be used. If the imputed date is for an AE start date and is in the same year and month as but after the last dose date + 30 days, then the last dose date + 30 days will be used.

If the imputed date is for an AE end date and is after the death date, the date of death will be used, or if the imputed AE end date is before the AE start date, the AE start date will be used.

### STATISTICAL METHODS OF ANALYSIS 9

### 9.1 **General Principles**

Descriptive statistics will be used to summarize baseline demographic and disease characteristics, study drug administration, efficacy and safety outcomes. Descriptive summaries of discrete data will present the sample size and the incidence as a frequency and as a percentage. Descriptive summaries of continuous data will present

Acerta Pharma 

Statistical Analysis Plan


the sample size, group mean, standard deviation (SD), median, and range. Confidence intervals (CIs) may be included as appropriate.

Summary tables will be presented by disease types: CLL/SLL, MCL, WM, FL, GCB DLBCL, MM, non-GCB DLBCL, RICHTER's and Other (include unclassifiable DLBCL, double hit lymphoma, FL with transformation, mediastinal DLBCL, mediastinal gray zone lymphoma, non-hodgkin's lymphoma [NHL], non-mediastinal gray zone lymphoma, red pulp small B-cell lymphoma, triple hit high grade NHL, hodgkin's lymphoma, marginal zone lymphoma), unless otherwise stated.

### 9.2 **Subject Accountability**

Subject disposition will be summarized for all treated subjects including the following information:

- Subject status on acalabrutinib and pembrolizumab
- Count and reason separately for acalabrutinib and pembrolizumab discontinuation
- Subject status for the study
- Count and reason for study termination
- Time on study
- Number of death

### 9.3 **Important Protocol Deviations**

Important Protocol Deviations (IPDs) categories are defined and managed by the study team during the IPD reviews throughout the study before database lock. These definitions of IPD categories, sub-category codes and descriptions will be used during the course of the study. The final IPD list is used to produce the summary of IPDs table and the list of subjects with IPDs.

The listing of the final IPD will be provided.

Statistical Analysis Plan


### 9.4 **Baseline Data**

Summaries of demographics and baseline characteristics will be presented for subjects in the all treated population. For continuous variables, mean, standard deviation, median, minimum, and maximum will be provided. For categorical variables, number and percentage of subjects in each category will be summarized.

### 9.4.1 **Demographics**

- Sex (Male, Female)
- Age (continuous)
- Age category (≥ 65)
- **Ethnicity**
- Race

# 9.4.2 Baseline Characteristics

- Height (cm)
- Weight (kg)
- ECOG performance status at baseline
- Bulky disease (grouped as  $\geq 5$  and  $\geq 10$  cm)
- Baseline B-symptoms (weight loss, fever and night sweats)
- Baseline Rai stage (CLL/SLL)
- Baseline Ann Arbor stage

### 9.5 **Treatment and Medications**

# **Prior Anticancer Therapies**

A prior anticancer therapy is defined as a systemic therapy subjects received, either as a single or combination therapy, for the treatment of active corresponding target disease with a start and end date occurring before the date of first dose of study treatment. Therapies given as a consolidation or maintenance of a response or remission will not be considered as a separate regimen. The number of lines and type of prior therapy will be summarized according to each disease cohort.

Acerta Pharma 


# 9.5.2 Prior and Concomitant Medications Received for Indications Other than **Target Disease**

Data reported on concomitant CRF page will be used. Medications started or ended prior to first dose will be consider as prior treatment. Concomitant therapy is defined as all medications used on or after the first dose, through the treatment phase, and for 30 days following the last dose of study drug. Using this definition, a medication can be classified as both prior and concomitant. Start date and end date will be imputed based on the rules provided in Section 12.1. of the SAP. Medications with completely missing start and stop dates will be considered as concomitant medications.

Prior and concomitant medications other than antineoplastic agents or other systemic therapies after enrollment will be summarized by the World Health Organization (WHO) Drug Dictionary therapeutic class, pharmacological class, and preferred term by each disease area.

# 9.5.3 Exposure to Study Drug

Descriptive statistics (n, mean, standard deviation, median, and range) will be used to summarize regarding the number of acalabrutinib doses prescribed:

- Total number of doses taken
- Duration of exposure (the interval between first dose date and last dose date)
- Average daily dose (the ratio of total dose administered and treatment duration)
- Relative dose intensities (the ratio of average daily dose and prescribed doses)
- The number and timing of prescribed dose reductions and interruptions

Descriptive statistics (n, mean, standard deviation, median, and range) will be used to summarize regarding the number of acalabrutinib doses prescribed:

- Total number of doses taken
- Duration of exposure (the interval between first dose date and last dose date)
- Average dose per cycle (total dose administered per cycle)
- Relative dose intensities (the ratio of average daily dose and prescribed doses)
- The number and timing of prescribed dose reductions and interruptions •

9.6 **Analyses of Efficacy Endpoints** 

9.6.1 **Response Rate** 

9.6.1.1 **Definition** 

Acerta Pharma 


ORR will be defined as the proportion of subjects who achieve a response defined in Section 4.2 in protocol for different disease. For lymphoma, response means partial response (PR) or better, for WM subjects response means miner response (MR) or better, for subjects with MF, response including clinical improvement or better (clinical improvement, PR, or CR). Please refer to Protocol section 4.2 for the detail information and definition of the response.

# 9.6.1.2 Analysis Methods

The primary analysis of ORR will be conducted on the all treated population. A descriptive analysis will be done on for subgroups of subjects who receive acalabrutinib alone or the combination of acalabrutinib and pembrolizumab. ORR and the corresponding 90% and 95% two-sided CI calculated using exact method to the binomial distribution will be presented.

The number and proportion of subjects within each category of response as well as the associated 95% CIs will be presented. The proportion will be estimated by dividing the number of subjects within each category of response by the total number of subjects in the analysis population. Each subject will be counted within only one response group, with the best response during the study as the classification group.

In addition, for subjects with CLL/SLL in Parts 1 and 2, a response will be assessed according to Table 4-2, which reflects modified International Working Group response criteria (Hallek 2008) as recently updated (Cheson 2012) to include PRL. For the purpose of this analysis, lymphocytosis at a given timepoint will be defined as absolute lymphocyte count which is above normal limits and is not ≥ 50% decreased from baseline. For Part 3 subjects with MF, an additional analysis will evaluate response when defined as CR + PR only.

# 9.6.2 Duration of Response

The duration of overall response (DOR) defined as the interval from the first documentation of response to the earlier of the first documentation of definitive disease progression or death from any cause. Subjects who had the event after the start of subsequent therapy, or are progression-free and alive at the time of data cutoff, or have unknown status will be censored at the last tumor assessment on or before the start of subsequent therapy and data cut-off time. The censoring rules for DOR are summarized in Appendix 12.2. The summary of DOR including mean, minimum, maximum, Q1 and Q3 are provided for all the responders for each disease group.

Acerta Pharma 

**Statistical Analysis Plan** 


9.6.3 Progression-free Survival

Progression-free survival (PFS) is defined as the interval from the first dose date of acalabrutinib or pembrolizumab to the earlier of the first documentation of objective disease progression or death from any cause. Subjects who had the event after the start of subsequent therapy, or who are progression-free and alive at the time of data cutoff, or have unknown status will be censored at the time of their last disease assessment on or before the start of subsequent therapy and data cut-off. Subjects with no post baseline disease assessment will be censored on Day 1. The censoring rules for primary

and sensitivity analyses of PFS are summarized Appendix 14.4.

The summary of PFS including the mean, minimum, maximum, median, Q1 and Q3 are

provided for all the responders for each disease group.

Summary of K-M estimates of PFS and 95% CIs as proper for each disease group

9.6.4 Time to Next Treatment

Time-to-next treatment defined as the time from the first dose date of acalabrutinib or pembrolizumab to the start of the next treatment other than the study treatment.

Descriptive statistics will be presented.

The summary of time to next treatment including the mean, minimum, maximum, median, Q1 and Q3 are provided for all the responders who have the next treatment for

each disease group.

9.6.5 Overall Survival

The duration of OS will be measured from the time of first study drug administration until the date of death from any cause. Subjects who are known to be alive as of their last known status will be censored at their last date known to be alive. Subjects who are lost in follow-up will be censored at the date the subject is last known to have been alive.

The censoring rules for OS are summarized Appendix 14.5.

The summary of OS including the mean, minimum, maximum, median, Q1 and Q3 are

provided for all the responders for each disease group.

Summary of 24 months K-M estimates of probability of OS including min, max, median

and 95% CIs are provided for each group as well.

Acerta Pharma 

Statistical Analysis Plan


# 9.6.6 Analysis Methods

The analysis of DOR will be conducted on the subset of the All-treated Population who are defined as responder in protocol section 4.2. The analysis of PFS and OS will be conducted on the All-treated Population. The analysis of DOR, PFS, and OS will be estimated using the Kaplan-Meier (KM) method. KM estimates with 95% CIs will be calculated for event time quartiles, and event-free rates will be calculated at selected time points. In addition, the reason for censoring will be summarized for DOR, PFS and OS.

### 9.7 **Analyses Safety Endpoints**

Safety analyses will be performed on the All-treated Population.

### 9.7.1 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA) will be used to code all AEs to a system organ class and a preferred term. The severity of the AE will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 or higher. Drug-related AEs are those assessed by investigator as related.

Treatment-emergent AEs are defined as those events that occur (actual or imputed start date) on or after the first dose of study drug, through the treatment phase, and within 30 days following the last dose of study drug.

Treatment-emergent AEs will be summarized by system organ class and preferred terms in descending order of frequency, by NCI toxicity grade and by relationship to study drug. The same summary will be provided for serious treatment-emergent AEs and drugrelated serious treatment-emergent AEs, treatment-emergent AEs leading to treatment discontinuation, dose reductions and dose withheld.

Death information is reported in the study exit CRF for all deaths. Incidences of deaths are to be reported, along with the primary cause of death.

AE by subject listing and death listing will be provided.

Acerta Pharma 

Statistical Analysis Plan


9.7.2 Laboratory Test Results

Laboratory data of hematology, serum chemistry up to 30 days after last dose or the

safety follow-up visit date, whichever is later, will be reported in SI units. Applicable

laboratory results will be graded according to CTCAE Version 4.03 or higher. Generic

normal ranges will be applied whenever reference ranges are not available.

Shift from baseline to the worst grade during the treatment will be provided as shift

tables for selected parameters. Figures of changes in selected parameters will be plotted

overtime as appropriate.

Urinalysis data will be summarized as appropriate.

By subject lab listing will be provided per each disease group.

9.7.3 Vital Signs

Summary statistics (mean, standard deviation, median, and range) will be produced for

vital signs at baseline, maximum, change from baseline to maximum, last value, and

change from baseline to last value.

In order to be included in the table, a subject must have both a baseline value and a

value for the given post-baseline time point.

By subject lab listing will be provided per each disease group.

9.7.4 ECOG Performance Status

Change of ECOG from baseline to the worst score during the treatment will be provided

as shift tables.

By subject ECOG listing will be provided per each disease group.

9.7.5 Physical Examinations

Physical examination data collected at screening and post-treatment will be

summarized. Descriptive statistics will be calculated for each parameters.

By subject physical examination listing will be provided per each disease group.

10 CHANGES FROM PROTOCOL-SPECIFIED ANALYSES

Acerta Pharma 


There is no major change from protocol-specified analyses.

# 11 LITERATURE CITATIONS / REFERENCES

Byrd JC, Harrington B, O'Brien S, et al. Acalabrutinib (ACP-196) in relapsed chronic lymphocytic leukemia. NEJM 2016;374:323-332.

Cheson BD, Pfistner B, Juweid ME, et al. Revised response criteria for malignant lymphoma. J Clin Oncol 2007; 25:579-586.

Cheson BD, Fisher RI, Barrington SF, et al. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol 2014;32:3059-3067.

Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0, USDHHS, NIH, NCI; publish date May 28, 2009 (v4.03: June 14, 2010).

FDA Drug Safety Communication 2012. Guidance for Industry and Investigators: Safety Reporting Requirements for INDs and BA/BE Studies (December 2012). Available at: http://www.fda.gov/downloads/Drugs/.../Guidances/UCM227351.pdf, accessed on: 13May2017.


### 12 **APPENDICES**

### 12.1 Study day

The study day will be calculated in reference to the date of first dose date. Study Day 1 is defined as the date of first dose of any study drug. For assessments that occur on or after first dose date, study day is defined as (date of assessment – date of first dose +

1). For assessments that occur prior to first dose date, study day is defined as (date of assessment – date of first dose). There is no Study Day 0.

### 12.2 **Censoring Rules for Duration of Response**

| Situation | Outcome | Date | Event Description/<br>Censoring Reason |
|---|---|---|---|
| Progression documented between scheduled visits on or before receiving subsequent anticancer therapy or data cutoff, whichever occurred first | Event | Earliest date of disease assessment documenting progression | PD |
| Death without documented PD on or before receiving subsequent anti-cancer therapy or data cutoff, whichever occurred first | Event | Date of Death | Death |
| New anti-cancer treatment Started before PD or death for subjects with or without documented PD or death and before data cutoff | Censored | Date of last adequate disease assessment prior to subsequent anti-cancer treatment | New anti-cancer<br>therapy |
| No documented PD or death at the time of data cutoff and subject not received subsequent anti-cancer therapy or subsequent anti-cancer therapy start date after the data cutoff | Censored | Date of last<br>adequate<br>disease<br>assessment on<br>or before data<br>cutoff | Data cutoff |
| Withdrew consent before documented PD or death | Censored | Date of last<br>adequate<br>disease<br>assessment | Withdrew consent |
| Lost to follow-up before documented PD or death | Censored | Date of last adequate disease assessment | Lost to follow-up |


### **Censoring Rules for Progression-free Survival** 12.3

| Situation | Outcome | Date | Event Description/<br>Censoring Reason |
|---|---|---|---|
| Progression documented between scheduled visits on or before receiving subsequent anticancer therapy or data cutoff, whichever occurred first | Event | Earliest date of disease assessment documenting progression | PD |
| Death without documented PD on or before receiving subsequent anti-cancer therapy or data cutoff, whichever occurred first | Event | Date of Death | Death |
| death before first adequate disease assessment | Event | Date of Death | Death |
| New anti-cancer treatment Started before PD or death for subjects with or without documented PD or death and before data cutoff | Censored | Date of last adequate disease assessment prior to subsequent anti-cancer treatment | New anti-cancer<br>Therapy |
| No documented PD or death at the time of data cutoff and subject not received subsequent anti-cancer therapy or subsequent anti-cancer therapy start date after the data cutoff | Censored | Date of last<br>adequate<br>disease<br>assessment on<br>or before data<br>cutoff | Data cutoff |
| Withdrew consent before documented PD or death | Censored | Date of last<br>adequate<br>disease<br>assessment | Withdrew consent |
| Lost to follow-up before documented PD or death | Censored | Date of last adequate disease assessment | Lost to follow-up |
| No post-baseline adequate disease assessments | Censored | Date of first<br>dose | No post-baseline adequate disease assessments |
| No baseline disease assessments | Censored | Date of first dose | No baseline disease assessment |


### **Censoring Rules for Overall Survival** 12.4

| Situation | Outcome | Date | Event Description/<br>Censoring Reason |
|---|---|---|---|
| Death on or before data cutoff | Event | Date of death | Death |
| Death or alive on or after data cutoff | Censored | Date of data cutoff | Data cutoff |
| Withdrew consent prior to data cutoff | Censored | Date of<br>discontinuation<br>from study<br>participation as<br>reported on<br>study exit CRF | Withdrew consent |
| Lost to follow-up prior to data cutoff | Censored | Date subject last known to be alive | Lost to follow-up |
| Survival status unknown on or after data cutoff | Censored | Date subject last known to be alive | Continue on study |